CLINICAL TRIAL: NCT01105221
Title: Acupuncture for Dry Eye: a Multicenter Randomized Controlled Trial With Active Comparison Intervention (Artificial Tear Drop) Using a Mixed Method Approach
Brief Title: Acupuncture for Dry Eye
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Korea Institute of Oriental Medicine (Other Government)
Collaborators: DongGuk University (Other); DONGSHIN University Oriental Hospital (Unknown)
Responsible Party: Kim, Ki-ok/ President of KIOM, Korea Institute of Oriental Medicine (KIOM)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KI1001
Record Dates: First submitted 2010-04-13; First posted 2010-04-16 (Estimated); Last update posted 2011-01-10 (Estimated); Status verified 2010-04

CONDITIONS: Dry Eye
Keywords: Acupuncture; Dry eye; Artificial tear drop; Mixed method approach; Qualitative study; Cost effectiveness analysis; Tear cytokine analysis
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Acupuncture (Experimental)
  Interventions: Device: Acupuncture
- Artificial tear drop (Active Comparator)
  Interventions: Drug: Refresh Plus

INTERVENTIONS:
Device: Acupuncture — Participants, allocated to this group, will have twelve times of acupuncture treatment in four weeks. Seventeen acupuncture points, which are both BL2, GB14, TE23, Ex1, ST1, GB20, LI4, LI11 and single GV23, will be selected and disposable 0.20*30mm acupuncture needles(Dongbang Co., Korea) will be inserted on these points. Strong 'deqi' sensation will be induced by twisting acupuncture needles and retained for 20 minutes before removed.
  Arms: Acupuncture
Drug: Refresh Plus — Participants, allocated to this group, will be offered preservative-free and single-use Refresh plus (Sodium carboxymethylcellulose). They should use artificial tear in both eyes at least once a day for four weeks.
  Other Names: Brand name: ALLERGAN
  Arms: Artificial tear drop

SUMMARY:
The purpose of this study is to assess whether acupuncture is more effective than artificial tear drop in the treatment of dry eye.

DETAILED DESCRIPTION:
Dry eye is one of the common diseases in ophthalmology. It affects not only patients' daily activities such as reading, carrying out professional work, using the computer, watching television, and driving, but also bodily health conditions such as bodily pain, discomfort and lower energy and vitality.

Currently, artificial tears are easily subscribed or used in the shape of OTC drugs. However, preservatives in artificial tears may exacerbate ocular surface inflammation and the safety of anti-inflammatory treatment is not well established.

Acupuncture, one of the most popular CAM interventions, showed some favourable effects over artificial tears for dry eye in several randomised controlled trials (RCTs). The evidence obtained from these trials is quite limited because all of these RCTs were conducted under high risk of biases. Therefore, well-designed RCTs are needed to establish the efficacy of acupuncture for dry eye.

In a clinical trial, cost-effectiveness and qualitative researches can be carried out parallely. Through this kind of mixed method approaches, various compartments, consisting acupuncture treatment effects are able to be revealed totally.

In this context, the investigators designed a multi-center randomized controlled trial, comparing acupuncture treatment and artificial tear drop with immunoassay for the change of tear cytokine concentration, cost effectiveness study and qualitative research in a mixed method approach.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have had dry eye syndromes in single eye or in both eyes (ICD-10 : H04.1). He or she must have both of the conditions below:

  1. Patients who have dry eye symptoms such as itching, ocular foreign body sensation, ocular burning, ocular pain, ocular dryness, blurred vision, sensation of photophobia, ocular redness, sensation of tearing
  2. Patients whose tear film break-up time is below 10 seconds and Schirmer I test results is below 10mm/5sec.

Exclusion Criteria:

* Patients who have defects of the eyelid or eyelashes
* Acute infection of the eyelid, eyeball or eye accessories
* Stevens-Johnson syndrome
* Vitamin A deficiency
* Eye or accessory defects due to external injuries
* A past history of surgical operation related to the eye in last three months
* Punctual occlusion
* Current usage of contact lenses
* Sequelae of facial palsy,
* Current usage of anti-inflammatory eye drops in the last two weeks
* Pregnancy
* Using history of traditional medicinal treatment such as acupuncture, moxibustion and herbal medicine in the last one month

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2010-04; Primary Completion 2010-11 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Ocular Surface Disease Index (OSDI) | Up to 13 weeks
  This questionnaire is a 12-item instrument for ocular irritation and impact on visual function in dry eye sufferers. It can provide quantifiable results of dry eye symptom frequency and vision-related functioning. Korean version of the OSDI questionnaire will be used. Follow up measurement will be assessed after 4, 5, 9 and 13 weeks from the first visit.

SECONDARY OUTCOMES:
Visual analogue scale (VAS) for self-assessment of ocular discomfort | Up to 13 weeks
  Self-reports on ocular symptoms concomitant with dry eye, such conditions as ocular itching, foreign body sensation, burning, pain and dryness as well as for blurred vision, sensation of photophobia, ocular redness and sensation of tearing. Follow up measurement will be assessed after 4, 5, 9 and 13 weeks from the first visit.
Schirmer I test with anaesthesia | Up to 13 weeks
  This ia a method for checking basic tear secretion. Schirmer test paper (Color Bar™ Eagle Vision, USA) will be inserted on the lateral third of the lower eyelid with the participant's eye closed for five minutes. Follow up measurement will be assessed after 5 weeks and 13 weeks from the first visit.
Tear Film Break Up Time (BUT) | Up to 13 weeks
  This is a method for observing tear film stability. Sodium fluorescein (2.5%) will be instilled in both eyes and the tear break-up time (the interval between the last complete blink and the first appearance of a dry spot or disruption in the tear film) will be measured. Follow up measurement will be assessed after 5 weeks and 13 weeks from the first visit.
General Assessment by acupuncture practitioner and participants | Up to 5 weeks
  Practitioners and participants will evaluate the improvement of ocular symptoms after treatment. They can chose one of the following 5 grades: Excellent, Good, Fair, Poor and Aggravation.
Self reports about experiences of using other dry eye-related treatments after the end of each intervention. | Up to 13 weeks
  For cost-effective analysis, all experience of using other dry eye-related treatments after the end of each intervention should be reported by participants. It contains frequency of hospital visit and treatments methods. Follow up measurement will be assessed after 9, 13 weeks from the first visit.
Quality of life (QOL) | Up to 13 weeks
  One questionaire for QOL, related to dry eye, is asked. Follow up measurement will be assessed after 4, 5, 9 and 13 weeks from the first visit.
Case reports on adverse events for the evaluation of safety | Up to 13 weeks
  Adverse events, adverse acupuncture or artificial tear drop reaction, serious and unexpected adverse acupuncture or artificial tear drop reaction and serious adverse event will be reported by participants and checked by practioners in every visit. Number of participants with adverse events will also be recorded.
Qualitative analysis (additional study) | Up to 13 weeks
  Questionaires with open-ended question about personal experiences for dry eye, acupuncture treatment and usage of artificial tear drop will be distributed to every participant of both group. Follow up measurement will be assessed after 4 and 13 weeks from the first visit.
Cost-effectiveness analysis between acupuncture and artificial tear drop treatment (additional study) | Up to 13 weeks
  Cost-effectiveness of acupucnture will be analyzed using Ocular Surface Disease Index (OSDI) variable, comparing the cost of artificial tear drops. the Cost which all participants will use for dry eye during the trial period, will be recorded in every visit.

CONTACTS AND LOCATIONS:
Overall Officials: Sun-Mi Choi, Dr, Principal Investigator — Korea Institute of Oriental Medicine
Locations (3):
- South Korea (3):
  - Clinical Research Center of DongGuk Univ. Internaltional Hospital, Goyang-si, Gyeonggi-do
  - Clinical Research Center of Korea Institute of Oriental Medicine, Daejeon
  - Clinical Research Center of DongShin Univ. Oriental Hospital, Gwangju

REFERENCES:
- [Derived] Kim TH, Kang JW, Kim KH, Kang KW, Shin MS, Jung SY, Kim AR, Jung HJ, Choi JB, Hong KE, Lee SD, Choi SM. Acupuncture for the treatment of dry eye: a multicenter randomised controlled trial with active comparison intervention (artificial teardrops). PLoS One. 2012;7(5):e36638. doi: 10.1371/journal.pone.0036638. Epub 2012 May 17. PMID 22615787
- [Derived] Kim TH, Kang JW, Kim KH, Kang KW, Shin MS, Jung SY, Kim AR, Jung HJ, Lee SD, Choi JB, Choi SM. Acupuncture for dry eye: a multicentre randomised controlled trial with active comparison intervention (artificial tear drop) using a mixed method approach protocol. Trials. 2010 Nov 16;11:107. doi: 10.1186/1745-6215-11-107. PMID 21078194